CLINICAL TRIAL: NCT03756961
Title: Effects of an Opioid Sparing Care Pathway for Patients Undergoing Obesity Surgery
Brief Title: Effects of an Opioid Free/Sparing Care Pathway for Patients Undergoing Obesity Surgery
Acronym: OS-PCC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OS-PCC-2017; 2017-003830-97 (EudraCT Number)
Record Dates: First submitted 2018-10-22; First posted 2018-11-28 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-11

CONDITIONS: Obesity; Pain, Postoperative
Keywords: opioids; bariatric surgery; anesthesia; opioid-free; person-centred care; recovery; TENS; pain
MeSH Terms: conditions — Obesity; Pain, Postoperative; Pain | interventions — Dexmedetomidine; Clinical Trials, Phase II as Topic; Esketamine; Ketamine; Lidocaine; Transcutaneous Electric Nerve Stimulation; Remifentanil; Desflurane; Propofol; Oxycodone

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, non-blinded, non-commercial multi centre study. The intervention is divided into 2 phases, and the two phases will primarily be analysed separately (i.e., between the control group and intervention Phase 1 and between the control group and intervention Phase 2)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): Control group: The patients receive the routine based anesthesiological treatment during bariatric surgery (Gastric By-Pass or Sleeve Gastrectomy). It consists of:
  General anesthesia induction: TCI Remifentanil Cpt 6 ng/ml/ Cp 3.2 ng/m, Propofol 1.5-2 mg/kg iv, Desflurane/Sevuflurane MAC (0.6-0.8).
  Maintained by Desflurane MAC (0.6-0.8) adjusted via BIS (40-60) and Remifentanil Cp 4-10 ng/ml.
  Post-operative pain management: Oxycodone 2.5 mg iv if the pain is rated by patient NRS ≧3. Paracetamol 1 g/6 h and Diclofenac 80 mg/24 h.
  Interventions: Drug: Remifentanil; Drug: Desflurane; Drug: Propofol; Drug: Oxycodone
- Intervention (Experimental): Induction: Dexmedetomidine 0.2 micrograms/kg/h iv 5 min+16 mcg, Esketamine 0.1mg/kg + Propofol 1.5-2 mg/kg iv, Desflurane/Sevuflurane MAC (0.6-0.8).
  Maintained by Desflurane/Sevuflurane MAC (0.6-0.8) BIS (40-60), Dexmedetomidine 0.2 micrograms/kg/h, Esketamine 0.1-0.3mg/kg/h och 0.1 mg/kg in case of hypertension. End of surgery, Lidocaine 1 mg/kg iv (max 4 mg/kg /4 h), Midazolam 0.5mg
  Post-operative: Dexmedetomidine (0.1-0.2 micrograms/kg/h up to 4 h post-operative). If the pain is rated NRS ≧3: Transcutaneous Nerve Stimulation (TENS) with high intensive 40-50 mA for 1 minute, if the patient still NRS ≧3, the TENS treatment is repeated one more time. If pain NRS ≧3 after two treatments with TENS: Esketamine 0.1mg/kg iv + Lidocaine 0.5 mg/kg iv (max 4 mg/kg /4 h) If pain NRS still ≧3 within 30 minutes after both TENS and Esketamine/Lidocaine, 2.5 mg Oxycodone iv until NRS < 3. Perioperative and at discharge, PCC will be used for the the intervention (Phase 2 patients)
  Interventions: Drug: Dexmedetomidine; Behavioral: Person-centred care (PCC); Drug: Esketamine; Drug: Lidocaine; Device: Transcutaneous Nerve Stimulation (TENS); Drug: Desflurane; Drug: Propofol

INTERVENTIONS:
Drug: Dexmedetomidine — The intervention group will obtain the pharmacological treatment during both perioperative. Pharmacological treatment in the intervention group differs solely from the patients in the control group by replacing opioids with the following non-opioid treatment:
  Other Names: Dexdor
  Arms: Intervention
Behavioral: Person-centred care (PCC) — The intervention tests non-pharmacological interventions compared to conventional treatment, supplemented by an evidenced-based Person-centred care PCC approach throughout the continuum of the perioperative and until 4 weeks after discharge. This will be part of patients in Phase 2
  Other Names: Phase 2
  Arms: Intervention
Drug: Esketamine — The intervention group will obtain the pharmacological treatment perioperatively. Pharmacological treatment in the intervention group differs solely from the patients in the control group by replacing opioids with the following non-opioid treatment:
  Other Names: Ketanest
  Arms: Intervention
Drug: Lidocaine — The intervention group will obtain the pharmacological treatment perioperatively. Pharmacological treatment in the intervention group differs solely from the patients in the control group by replacing opioids with the following non-opioid treatment.
  Other Names: Xylocaine
  Arms: Intervention
Device: Transcutaneous Nerve Stimulation (TENS) — The intervention group will obtain non-pharmacological treatment by TENS during the entire hospital stay (both perioperative and post-operative) until discharge.
  Other Names: TENS
  Arms: Intervention
Drug: Remifentanil — The control group receives general anesthesia with Remifentanil as the routine opioid drug during general anesthesia.
  Other Names: Ultiva
  Arms: Control
Drug: Desflurane — The patient receives general anesthesia with Desflurane/ or Sevoflurane as the routine volatile anesthetic during general anesthesia
  Other Names: Desfluran
Drug: Propofol — The patient receives general anesthesia with Propofol as the routine induction anaesthetic during general anesthesia
Drug: Oxycodone — The control group receives Oxycodone as the routine pain management drug post-operative.
  Arms: Control

SUMMARY:
The opioid consumption has exploded in the western world, and for some patient populations such as obese patients, patients with sleep apnoea or patients undergoing cancer treatment, opioid-sparing/ opioid-free strategies could have positive effects on outcomes. Studies suggest that opioids could have opioid-induced immunosuppression, induce chronic post-operative pain syndrome and hyperalgesia in addition to the more well-known side effects such as respiratory depression, nausea, bladder, and bowel dysfunction. Hence, new studies are needed on the impact of person-centered care programs that combine pharmaceutical and non-pharmaceutical strategies to reduce the adverse short and long-term effects of opioid therapy.

The overall aim is to evaluate the short-, medium- and long-term effects of opioid-free care pathways with or without person-centred care compared to conventional opioid-based treatment in patients undergoing obesity surgery.

Specific aims

1. Determine the effects of opioid-free care with or without person-centred care compared with conventional opioid-based general anaesthesia on the cognitive and physical quality of recovery after surgery up to 24 months after surgery (short-term: postoperative to discharge, medium-term: 14 days, 3 months, long-term: 6 months, 12 months and 24 months).
2. Describe the clinical monitoring trend regarding nociceptive response intraoperatively between opioid-free and conventional care.
3. Map the impact of opioid-free anaesthesia (with and without person-centred care) on the usage of opioids up to 24 months after hospital discharge.
4. Explore the patients' experience of quality of life, economic evaluations, self-efficacy and recovery after surgery in opioid-free care with or without person-centred care during the first year post-surgery.

The aims will be evaluated by a prospective, randomized, non-blinded, non-commercial multi-centre study (Nov 2018-Dec 2022) approved by the Swedish Medicines Agency (EU-CT 2023-505934-86-00) and the ethical review board (DNR 1006-17).

DETAILED DESCRIPTION:
Aim To evaluate the effects of opioid sparing care pathways compared to conventional opioid-based treatment for pain relief, opioid consumption, recovery after surgery, self-efficacy and health economy in patients undergoing obesity surgery. The aim will be investigated by a prospective, randomized, non-blinded, non-commercial multi-centre study(Nov 2018-Dec 2022), approved by the Swedish Medicines Agency (EU-CT 2023-505934-86-00) and the ethical review board (DNR 1006-17).

Hypothesis 1. An opioid-free care pathway provides non-inferior pain relief as the conventional care with opioids during the post-operative phase.

Primary endpoints: Determine the quality of recovery after surgery

1. No difference in pain (NRS pain (0-10)) between opioid-free intervention with or without (Phase 1 & 2) person-centred care and conventional treatment (control group) during the postoperative phase until discharge to the surgical ward.

Secondary endpoints:

An opioid-sparing treatment provides improved combined outcomes (composite score) consisting of 1) Self-Efficacy, 2) Postoperative Quality of Recovery Scale (PQRS), hospital readmission, or death at 3 months compared to conventional treatment.

An opioid-sparing treatment results in reduced opioid consumption during the peri- and postoperative period until discharge to the ward compared to conventional treatment.

An opioid-sparing treatment results in reduced opioid consumption throughout the hospital stay compared to conventional treatment.

An opioid-sparing treatment results in decreased pain experience according to the Numeric Rating Scale (NRS) at 3 months and 6 months compared to conventional treatment.

An opioid-sparing treatment leads to earlier recovery after surgery measured with PQRS compared to conventional treatment postoperatively (20 minutes, 40 minutes), during hospitalization (24-72 hours), and thereafter (14 days, 30 days, 3 months, 6 months, 12 months, and 24 months).

An opioid-sparing treatment increases confidence in coping with unexpected events measured with the General Self-Efficacy Scale compared to conventional treatment after the in-hospital period (3 months, 6 months, 12 months, 24 months).

An opioid-sparing treatment improves quality of life measured with RAND-36 and EQ5D compared to conventional treatment after the in-hospital period (3 months, 6 months, 12 months, 24 months)

An opioid-sparing treatment results in equivalent length of hospital stay compared to conventional treatment during the in-hospital period.

Mapping of long-term prescription of analgesic drugs. Does an opioid-sparing treatment impact the long-term use of analgesic medications.

Explorative endpoints:

Describe the intraoperative nociception level between opioid-free anaesthesia and conventional anaesthesia using the Medasense PMD-200 (NOL) monitor.

Economic evaluation: Performing cost-utility analysis/ cost-effectiveness analyses.

Power Pain: To determine noninferiority with a power of 0.8 (i.e., the probability of > 0.8 for the lower limit of a two-sided 95% confidence interval (using Fisher's nonparametric permutation test)), the difference of change in pain using the NRS from arrival to the recovery unit after surgery to discharge from the recovery unit will be used. Forty-three patients are required in each group and phase, with an SD for the change in the NRS estimated to be 1.62 from a small pilot study (noninferiority margin -1.0). The estimated change was assumed to be equal in the groups. To compensate for a potential interruption in the study or dropouts, we chose to include 55 patients in Intervention Phase 1, 55 patients in Intervention Phase 2 and a total of 110 patients in the control group (to follow intervention Phases 1 and 2, each 55 patients).

Recovery after surgery: To detect an overall difference in the quality of recovery between groups over the entire study length, with a power of 0.8 and P < 0.05 and taking into consideration a dropout of over 30% as seen in other studies using the PQRS, we need to include at least 30 patients in each group 26.

The control group will receive usual care and treatment according to the hospital's routines, where pain relief is obtained with opioids postoperatively. Pharmacological treatment in the intervention group differs solely from the patients in the usual group by replacing opioids with the following nonopioid perioperative treatment: dexmedetomidine, esketamine, lidocaine and TENS (for exact dosing, please visit EU-CT 2023-505934-86-00). Postoperative patient-controlled pain treatment with high-intensity/high-frequency TENS is used if the patient perceives pain over NRS ≧ 3 postoperatively and during remaining hospitalisation.

Intervention Phase 1 tests the pharmacological and non-pharmacological interventions (TENS) compared to the control group that receives standard care with opioids intra- and postoperatively. Phase 2 intervention that follows after completion of Phase 1 intervention tests the pharmacological and nonpharmacological interventions compared to conventional treatment, supplemented by an evidenced-based PCC approach throughout the continuum of postoperative care.

The two phases will primarily be analysed separately (i.e., between the control group and intervention Phase 1 and between the control group and intervention Phase 2).

ELIGIBILITY:
Inclusion Criteria:

-Patients ≥18 years planned to undergo laparoscopic obesity surgery (GBP alt Sleeve surgery) at the selected site.

Exclusion Criteria:

* ASA> III
* Cardiovascular disease with bradycardia (<50 bpm)
* Serious liver disease failure
* Insufficient knowledge of the Swedish language
* Serious untreated psychiatric disease
* Neurocognitive dysfunction
* Pregnancy
* Women of childbearing age without contraception
* Malignant disease with expected short survival
* Patients treated with opioids for chronic pain
* Substance abuse
* Hypersensitivity to Oxycodone, Esketamine, Dexmedetomidine, and Lidocaine
* Pacemaker or ICD
* Inability to fill in questionnaires
* Decline participation,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference in post-operative pain from admission to the post-anesthesia care unit (PACO) to discharge from the PACO unit to the surgical ward. | From date of randomization, difference in NRS will be assessed as the change in NRS from arrival (20 minutes after arrival) to the post-anesthesia care unit(PACU) after the surgery, to the time of discharge ( 4 hour) from the PACU to the surgical ward
  Post-operative phase until discharge to the surgical ward. Pain assessed according to change in NRS (numeric rating scale). NRS (numeric rating scale for pain), (ranging from 0-10, "no pain" vs. "worst imagined pain").

SECONDARY OUTCOMES:
Recovery after surgery | (20 min, 40 min), during hospitalization (24 hours-72 hours) and afterwards (14 days, 30 days, three months, six months, 12 months and 24 months)
  Investigating recovery after surgery measured with the The Post-operative Quality of Recovery Scale (PostopQRS) compared with conventional postoperative therapy.
  PostopQRS: Is a validated 5-dimensional instrument (Physiology, Nociception, Emotion, Cognition, ADL) in addition to questions about patient satisfaction.
  The scoring of recovery is 'return to baseline values or better' which requires a change score ≥ 0 for each question. The postoperative value for each test ( Cognition has a 2 scale tolerance due to day-to-day variation) is subtracted from the baseline value, and if no difference, then the patient is recovered.
Average opioid consumption perioperative | From the start of the Peri-operative phase (start of surgery) until discharge from hospital ( index stay), up to 24 months post-discharge
  Investigating opioid consumption during the peri- and post-operative care period compared with conventional treatment until discharge from the hospital and up to 24 months discharge.
Length of hospital stay | Indexed length of hospital day will be calculated in days/hours). Estimated stay is 2 days
  Length of indexed hospital stays calculated as the mean length in days from admission to discharge
Change in general Self-Efficacy | 3 months, six months, 12 months, 24 months.
  Investigating patient change in self-efficacy, measured with the General Self-Efficacy Scale (GSES). GSES is a validated questionnaire that contains 10 questions about the person's experiences of trust in his / her ability to handle difficult situations. The patient is asked to estimate his ability on a 4-point scale (1 not true) to 4 (true).
  The 10 answers are summed and a mean is calculated. Higher scores are better.
Change in Quality of Life | (3 months, six months, 12 months, 24 months)
  Investigating the quality of life measured with the RAND-36
  RAND-36: The RAND-36 is a health-related quality of life (HRQoL) It is comprised of 36 items assessing eight areas: physical functioning, role limitations caused by physical health problems, role limitations caused by emotional problems, social functioning, emotional well-being, energy/fatigue, pain, and general health perceptions.
  Each item is scored 0-100, and are than summarized. 0 is low, 100 is the highest score to get.
Exploring patient experience | 2 weeks after hospital discharge
  Investigating patient experience and satisfaction during the hospital stay, measured with the PPE-15, a 15 item questionnaire. The PPE15 is a validated short version of The Picker Care experience survey (40 item).
  Each item has response alternatives ranging from no problem, some problem, problem. Each response is coded either as "a problem" ( problem, some problem) or as "no problem". Problem is scored as=1, no problem=0. The mean is calculated both on item level and as a total score.
Change in health status | (3 months, six months, 12 months, 24 months)
  Investigating the change in health status measured with the EuroQol 5 dimension (EQ5D).
  EQ-5D is a standardized instrument for measuring generic health status, covering five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
  Each dimension has 3 responses: no problems, some problems, and extreme problems. This response results into a number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state'.
Unplanned re-admission | From time of surgery up until 24 months post-surgery
  Investigating re-admission (un-planned) between groups.
Mortality | From time of surgery up until 24 months post-surgery
  Investigating mortality rate between groups.

OTHER OUTCOMES:
Economic evaluation | During hospital stay and up to 24 months
  Performing cost-utility analysis/ cost-effectiveness

CONTACTS AND LOCATIONS:
Overall Officials: Sven-Egron Thörn, MD, PhD, Principal Investigator — Göteborg University; Axel Wolf, RN, PhD, Professor, Study Chair — Göteborg University
Locations (2):
- Sweden (2):
  - Lindesberg Hospital, Lindesberg, Region Örebro
  - Sahlgrenska University hospital/ Östra hopsital, Gothenburg, VG

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Olausson A, Jildenstal P, Andrell P, Angelini E, Stenberg E, Wallenius V, Ohrstrom H, Thorn SE, Wolf A. Effects of an opioid-free care pathway vs. opioid-based standard care on postoperative pain and postoperative quality of recovery after laparoscopic bariatric surgery: A multicentre randomised controlled trial. Eur J Anaesthesiol. 2025 Aug 1;42(8):714-726. doi: 10.1097/EJA.0000000000002193. Epub 2025 May 14. PMID 40371564